CLINICAL TRIAL: NCT00034593
Title: A Phase 2 Trial of ALIMTA (Pemetrexed) Plus Gemcitabine in Locally Advanced or Metastatic Transitional Cell Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 4699; H3E-MC-JMEV
Record Dates: First submitted 2002-04-30; First posted 2002-05-01 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Urologic Neoplasms
Keywords: Bladder cancer; metastatic; transitional cell carcinoma of the urothelium
MeSH Terms: conditions — Urologic Neoplasms; Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: ALIMTA
Drug: gemcitabine

SUMMARY:
Definition: Patients with bladder cancer will be participating in this study for the treatment of abnormal cells in the bladder that have returned after initial treatment OR have moved to a new site in the body.

ELIGIBILITY:
Inclusion Criteria:

* You must have been diagnosed with bladder cancer that has recurred or moved to a new part of the body.
* You must have at least one tumor that can be physically measured or scanned by x-ray.
* You may not have had previous chemotherapy (drug) treatment OR you have had surgery followed by one chemotherapy treatment at least 4 months ago.

Exclusion Criteria:

* You may not have used an experimental medicine or device within the past month.
* Cancer that has spread to your brain.
* If you are unwilling or unable to take folic acid or vitamin B12 supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- Finland (3):
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Helsinki
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Pikonlinna
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Turku
- France (5):
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Bordeaux
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Lille
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Marseille
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Montpellier
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician.", Paris
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Homburg/Saar, Germany